CLINICAL TRIAL: NCT05580042
Title: An Open-Label, Single Arm, Phase I Study to Evaluate the Safety and Tolerability of AC-1101 Topical Gel in Patients with Granuloma Annulare
Brief Title: Study to Evaluate the Safety and Tolerability of AC-1101 Topical Gel in Patients with Granuloma Annulare
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-1101-GA-001
Record Dates: First submitted 2022-10-02; First posted 2022-10-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Granuloma Annulare
Keywords: Tofacitinib Topical Gel 2%; AC-1101 gel
MeSH Terms: conditions — Granuloma Annulare

STUDY DESIGN:
Intervention Model Description: patients with Granuloma Annulare
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Granuloma Annulare (Experimental): 4-week treatment and 2-week follow-up period (without treatment)
  Interventions: Drug: AC-1101

INTERVENTIONS:
Drug: AC-1101 — For each patient, once daily (QD)
  Other Names: Tofacitinib Topical Gel 2%; AC-1101 gel

SUMMARY:
Study AC-1101-GA-001 is an early phase open-label study with a 4-week treatment and 2-week follow-up period (without treatment) to assess the safety, tolerability, and efficacy of AC-1101 gel in patients with Granuloma Annulare.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older, male or female, will be enrolled.
2. Diagnosis of granuloma annulare with supportive skin biopsy (diagnostic shave biopsy or punch biopsy) or historical biopsy (a provided report would be sufficient and would not require to repeat the diagnostic biopsy). A biopsy at any point is sufficient. If a diagnostic biopsy has never been performed, one will be performed prior to enrollment in the study. Patients with both localized and generalized GA will be enrolled in the proposed study.
3. Other subtypes of GA, such as linear, perforating, and subcutaneous will be excluded from the study. If there is suspicion that GA is medication-induced, the patient will not be enrolled. GA in association with human immunodeficiency virus (HIV) or malignancy will be excluded.
4. Patients with 1-20% BSA of active Granuloma Annulare lesions will be enrolled.
5. Duration of active GA must be at least two years with no significant change in size or number of lesions in the 6 months prior to treatment as supported by a combination of record review and history/patient interview.
6. Patients who might be recalcitrant to or intolerant of conventional treatment, such as antibiotics (e.g., doxycycline or minocycline), triple antibiotic therapy of rifampin, ofloxacin, and minocycline, topical corticosteroids, topical calcineurin inhibitors, intralesional/intramuscular corticosteroid and/or phototherapy.
7. Adequate organ function and marrow function meaured at screening (Visit 1) and enrollment (Visit 2) as defined below:

   * Hemoglobin ≥ 12.0 g/dL for male and 10.5 g/dL for female;
   * Absolute neutrophil count ≥ 1,300 /µL;
   * Absolute lymphocytes: 1.0-4.0 x 109/L (1000-4000 cells/mm3) as the reference range;
   * Platelets ≥ 75,000/µL;
   * Total bilirubin ≤ 1.5 x upper normal limit;
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 x upper normal limit;
   * eGFR ≥ 60mL/min/1.73m2
8. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration.

   * Intra-uterine contraceptive device without hormone release system placed at least 4 weeks prior to study drug administration.
   * Male partner using condom with intravaginally applied spermicide started at least 21 days prior to study drug administration.
   * Sterile male partner (vasectomized since at least 6 months).
   * Barrier method of contraception: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, bilateral tubal occlusion, sexual abstinence (when this is in line with preferred and usual lifestyle). No combined hormonal contraceptive methods (such as most oral pills, rings or patches) are permitted.
9. Capable of consent: Able to read, understand, and sign the Informed Consent Form (ICF), answer the study questionnaires, communicate with the Investigator, and understand and comply with protocol requirements.
10. Patients must speak English.
11. Patients must have health insurance.

Exclusion Criteria:

1. Patients with active malignancy will not be permitted to enroll in the proposed study. Patients with a history of treated nonmelanoma skin cancer will be eligible to enroll.
2. Patients under treatment with biologics or other systemic immunosuppressive medications (e.g., methotrexate (MTX), mycophenolate) within the last 3 months.
3. Presence of any clinically significant abnormality at physical examination, clinically significant abnormal laboratory assessment or positive test for hepatitis B (HBs-Ag), hepatitis C (HCV-Ab), or HIV found during medical screening.
4. History of allergic reactions to tofacitinib or other related drugs, or to any excipient in the formulation.
5. Positive pregnancy test at screening. If a woman becomes pregnant during the study, she will stop the study medication and be removed from the study. She will be urged to follow up with her Primary Care Physician or obstetrician-gynecologist. The study doctors will ask to follow the pregnancy to its outcome.
6. Women of childbearing potential who are unable or unwilling to use birth control (oral pills, rings or patches are not permitted) while taking the medication.
7. Pregnant or breast-feeding women.
8. Current active smokers.
9. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving drug or device administration.
10. History of active tuberculosis or exposure to endemic areas within 8 weeks prior to QuantiFERON®-TB testing performed at screening.
11. Positive QuantiFERON®-TB indicating possible tuberculosis infection.
12. Immunization with a live attenuated vaccine within 1 month prior to dosing or planned vaccination during the study.
13. History of clinically significant opportunistic infection, e.g., invasive fungal infections or pneumocystis pneumonia.
14. Serious local infection, e.g., cellulitis, abscess, or systemic infection, e.g., septicemia, within 3 months prior to screening.
15. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis, such as Acetaminophen (2g in 24-hour period) because they are judged unlikely to affect the PK profile of the study drug or subject safety:

    1. Prescription medications within 14 days prior to the first dosing with the exception of on-going medications to treat existing comorbid disorders, as judged by the Investigator.
    2. Topical medications inlcuding antibiotics or corticosteriod applied to the designated treatment area.
    3. Depot injection or implant of any drug within 3 months prior to the first dosing.
    4. Any drugs known to significantly induce or inhibit hepatic drug metabolism via the CYP3A4 and CYP2C19 enzymes within 30 days prior to first dosing.
16. Fever associated with a symptomatic viral or bacterial infection, within 2 weeks prior to the first dosing.
17. Subjects with a personal history of significant coronary heart disease, heart failure, and/or cerebrovascular disease.
18. Any reason that, in the opinion of the Investigator, would prevent the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence and proportion of subjects with treatment emergent adverse events (TEAEs), AEs and serious adverse events (SAEs). | Up to 6 weeks
  Adverse events (AEs), Significant Adverse Events (SAEs), treatment emergent adverse events (TEAEs)
Number of subjects with abnormal vital signs | Up to 6 weeks
  Vital sign parameters will be analyzed including oral temperature, pulse rate, respiratory rate, and blood pressure.
Number of subjects with abnormal ECG | Up to 6 weeks
  ECGs will be obtained by using an automated ECG machine to measure PR, QRS, QT, and QTc intervals and calculates heart rate.
Number of subjects with abnormal hematology parameters | Up to 6 weeks
  Hematology parameters will be analyzed including platelet count, RBC count, hemoglobin, hematocrit, MCV, MCH, percent reticulocytes, WBC count, neutrophils, lymphocytes, monocytes, eosinophils and basophils.
Number of subjects with abnormal biochemistry parameters | Up to 6 weeks
  Biochemistry parameters will be analyzed including blood urea nitrogen (BUN), creatinine, glucose, phosphorus, calcium, phosphate, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transferase (GGT), alkaline phosphatase, creatine phosphokinase (CPK), total bilirubin, direct bilirubin, total protein, albumin to gloulin ratio, globulin, lipase, and Hemoglobin A1C..
Number of subjects with abnormal urinalysis parameters | Up to 6 weeks
  Urinalysis parameters will be analyzed including specific gravity, urine creatinine, phosphate and pregnancy test..
Change in skin irritation using Dermal Rating Scale (DRS) | Up to 4 weeks
  This is a 0-4 rating with 0 representing the best.

SECONDARY OUTCOMES:
Plasma concentration of AC-1101 | Day 1, Day 14, Day 42:Pre-dose; Day 28: Pre-dose, 2 through 24 hours post-dose
  Blood samples will be collected from patients from Visit 2 to Visit 5
Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration (AUC[0-t]) of AC-1101 | Day 1, Day 14, Day 42:Pre-dose; Day 28: Pre-dose, 2 through 24 hours post-dose
  Blood samples will be collected from patients from Visit 2 to Visit 5
Area under the plasma concentration-time curve from time 0 to extrapolated to infinity (AUC[0-infinity]) of AC-1101 | Day 1, Day 14, Day 42:Pre-dose; Day 28: Pre-dose, 2 through 24 hours post-dose
  Blood samples will be collected from patients from Visit 2 to Visit 5
Maximum observed plasma drug concentration (Cmax) of AC-1101 | Day 1, Day 14, Day 42:Pre-dose; Day 28: Pre-dose, 2 through 24 hours post-dose
  Blood samples will be collected from patients from Visit 2 to Visit 5
Time to maximum observed plasma drug concentration (Tmax) of AC-1101 | Day 1, Day 14, Day 42:Pre-dose; Day 28: Pre-dose, 2 through 24 hours post-dose
  Blood samples will be collected from patients from Visit 2 to Visit 5
Apparent terminal half-life (T1/2) of AC-1101 | Day 1, Day 14, Day 42:Pre-dose; Day 28: Pre-dose, 2 through 24 hours post-dose
  Blood samples will be collected from patients from Visit 2 to Visit 5

OTHER OUTCOMES:
Change in Patient Global Impression of Change in GA (PGIC-GA) | Up to 4 weeks
  This is a 1-5 rating with 1 representing the much improved.
Change in Dermatology Life Quality Index (DLQI) | Up to 4 weeks
  The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above. There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range form 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Change in Skindex-16 | Up to 4 weeks
  This is a patient quality of life survey using the skindex 16 survey form. The 16-item Skindex questionnaire is divided into three domains: questions related to the participant's symptoms (1-4), emotions (5-11), and functioning (12-16). Each question asks the participant to quantify how much a specific aspect of their skin condition bothered them in the week prior to administration of the Skindex-16. The questions are answered on a scale from 0 (no impact) to 6 (significant) with a total possible score ranging from 0 (best) to 96 (worst). Each item is then transformed to a linear scale from 0 to 100.
Change in GA-Investigator Global Assessment (GA-IGA) score for the treated GA lesions | Up to 4 weeks
  This is a 0-4 rating with 0 representing the clear.
Change in Granuloma Annulare Severity and Morphology Instrument (GASMI) activity score for the treated GA lesions | Up to 4 weeks
  The GASMI includes ten body regions, scored by inflammation (scores 1, 2, 4), induration (scores 1, 2, 3), and area (scores 1, 2, 3, 5, 7). The total score may vary from 30 (best) to 140 (worst).
Percent change in BSA of the treated GA lesions | Up to 4 weeks
Proportion of patients who have complete response (defined as no active disease clinically) and partial response | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Damsky, M.D., Ph.D., Principal Investigator — Yale Department of Dermatology
Locations (1):
- Yale Center for Clinical Investigation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No